CLINICAL TRIAL: NCT04330274
Title: Comparison of Different Amputation Levels in Terms of Balance Parameters and Plantar Pressure Distribution; Lower Extremity
Brief Title: Comparison of Different Amputation Levels
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.357
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2019-04

CONDITIONS: Amputee; Plantar Pressure Distrubution; Balance
Keywords: amputee,plantar pressure, balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Unilateral transtibial amputee
  Interventions: Other: Bipedal with open eyes; Other: Bipedal with closed eyes; Other: Bipedal with open eyes and with platform; Other: Bipedal with closed eyes and with platform
- Group 2: Unilateral transfemoral amputee
  Interventions: Other: Bipedal with open eyes; Other: Bipedal with closed eyes; Other: Bipedal with open eyes and with platform; Other: Bipedal with closed eyes and with platform

INTERVENTIONS:
Other: Bipedal with open eyes — Standing bipedal with open eyes on force platform
Other: Bipedal with closed eyes — Standing bipedal with closed eyes on force platform
Other: Bipedal with open eyes and with platform — Standing bipedal with open eyes and with platform under heel of prosthetic foot on force platform
Other: Bipedal with closed eyes and with platform — Standing bipedal with closed eyes and with platform under heel of prosthetic foot on force platform

SUMMARY:
Lower limb amputation is a factor that changes the individual's weight transfer, gait pattern, and trunk balance. This change plantar pressure distribution of both side and cause a series of problems to be exposed over time according to level of amputation. The aim of this study is to reveal the relationship between amputation level-postural balance and amputation level-plantar pressure distribution.

ELIGIBILITY:
Inclusion Criteria:

* Being unilateral transfemoral or transtibial amputee
* Have the level of perception to understand and apply the commands given
* Having sedantary life styles

Exclusion Criteria:

* Having a neurological or orthopedic disorder that may affect standing posture and balance
* The presence of pain that can affect standing posture and balance
* Visual impairment that impairs the gait pattern and balance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unilateral transtibial and transfemoral amputees
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of plantar pressure distrubution | Change from baseline plantar pressure distrubution at second 10, second 20 and second 30.
  Plantar pressure distrubution (mmHg/N) will be measured by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with open eyes
Measurement of plantar pressure distrubution | Change from baseline plantar pressure distrubution at second 10, second 20 and second 30.
  Plantar pressure distrubution (mmHg/N) will be measured by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with platform under heel
Determination of center of pressure | Change from baseline center of pressure at second 10, second 20 and second 30.
  Determination of center of pressure (cm) will be provided by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with open eyes
Determination of center of pressure | Change from baseline center of pressure at second 10, second 20 and second 30.
  Determination of center of pressure (cm) will be provided by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with platform under heel.
Measurement of plantar pressure distrubution | Change from baseline plantar pressure distrubution at second 10, second 20 and second 30.
  Plantar pressure distrubution (mmHg/N) will be measured by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with closed eyes
Measurement of plantar pressure distrubution | Change from baseline plantar pressure distrubution at second 10, second 20 and second 30.
  Plantar pressure distrubution (mmHg/N) will be measured by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal without platform under heel
Determination of center of pressure | Change from baseline center of pressure at second 10, second 20 and second 30.
  Determination of center of pressure (cm) will be provided by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal with closed eyes
Determination of center of pressure | Change from baseline center of pressure at second 10, second 20 and second 30.
  Determination of center of pressure (cm) will be provided by force platform (F-Scan 6.70 TekScan, Boston, MA) on bipedal without platform under heel.

CONTACTS AND LOCATIONS:
Overall Officials: yasar tatar, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jayakaran P, Johnson GM, Sullivan SJ. Postural control in response to altered sensory conditions in persons with dysvascular and traumatic transtibial amputation. Arch Phys Med Rehabil. 2015 Feb;96(2):331-9. doi: 10.1016/j.apmr.2014.09.037. Epub 2014 Oct 22. PMID 25450125
- [Background] Castro MP, Soares D, Mendes E, Machado L. Plantar pressures and ground reaction forces during walking of individuals with unilateral transfemoral amputation. PM R. 2014 Aug;6(8):698-707.e1. doi: 10.1016/j.pmrj.2014.01.019. Epub 2014 Jan 29. PMID 24487128
- [Background] Marks RM, Long JT, Exten EL. Gait abnormality following amputation in diabetic patients. Foot Ankle Clin. 2010 Sep;15(3):501-7. doi: 10.1016/j.fcl.2010.05.001. PMID 20682420
- [Background] Nolan L, Wit A, Dudzinski K, Lees A, Lake M, Wychowanski M. Adjustments in gait symmetry with walking speed in trans-femoral and trans-tibial amputees. Gait Posture. 2003 Apr;17(2):142-51. doi: 10.1016/s0966-6362(02)00066-8. PMID 12633775